CLINICAL TRIAL: NCT02248441
Title: Effect of Remote Ischemic Conditioning in Patients With Chronic Ischemic Heart Failure (CONDI-HF)
Brief Title: Effect of Remote Ischemic Conditioning in Patients With Chronic Ischemic Heart Failure
Acronym: CONDI-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEK: 1-10-72-173-14
Record Dates: First submitted 2014-09-02; First posted 2014-09-25 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2016-10

CONDITIONS: Chronic Systolic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily RIC (Experimental): Daily ischemic conditioning treatment
  Interventions: Other: Daily ischemic conditioning treatment

INTERVENTIONS:
Other: Daily ischemic conditioning treatment — RIC stimulus will be conducted as 4 x 5 minutes upper arm ischemia achieved by inflation of a blood pressure cuff to 200 mmHg and 5 minutes reperfusion between inflations. The procedure will be performed using the AutoRICTM (CellAegis Devices Inc., Toronto, Ontario, Canada).

SUMMARY:
The present study will evaluate whether treatment with daily remote ischemic conditioning for a 28±4-day period induces beneficial effects in subjects with and without chronic ischemic heart failure in terms of improved left ventricular contractile function and exercise capacity.

DETAILED DESCRIPTION:
Background Chronic heart failure (CHF) is a leading cause of morbidity and mortality throughout the world, and the incidence and prevalence are increasing as more patients survive their acute coronary syndrome. The disease is caused by abnormalities in cardiac structure or function leading to insufficient delivery of oxygen to the metabolizing tissues. These patients are often debilitated, require chronic medications, and many receive expensive device therapy to manage symptoms. Consequently, this has led to an increasing economic and health burden from heart failure.

CHF is the end-stage of a broad range of underlying cardiovascular diseases, but is most frequently caused by ischemic heart disease. Other contributory causes include hypertension, heart valve diseases, arrhythmias and cardiomyopathies, all resulting in myocardial tissue damage and loss of ventricular function. Activation of neurohormonal and inflammatory compensatory mechanisms lead to a vicious circle through adaptive metabolic and remodeling processes, eventually resulting in a progressive decline of cardiac function with significant morbidity and mortality.

Identification of the specific underlying cardiac condition is crucial for the therapeutic approach in patients suffering from CHF. While pharmacological treatment remains dominating, resynchronization therapy and surgical resection of non-contractile tissue are also increasingly being conducted. Despite the fact that activation of the inflammatory system greatly contributes to the remodeling process through initiation of myocardial fibrosis and hypertrophy, most clinical studies targeting inflammatory components have been discouraging.

Remote ischemic conditioning (RIC) by brief non-lethal episodes of ischemia in a remote organ or tissue (e.g. a limb) is a novel therapeutic method to achieve protection against ischemia-reperfusion injury in the target organ, e.g. the heart . In the clinical setting, RIC is most often performed by repeated episodes of limb ischemia achieved by intermittent inflation of a blood pressure cuff placed around the upper arm. In clinical randomized trials, RIC has been shown to reduce the amount of myocardial injury and improve long-term outcome in patients admitted with STEMI for primary percutaneous coronary intervention and patients undergoing cardiac surgery or elective coronary intervention.

RIC is a low-cost, simple and safe procedure that can easily be conducted using a standard blood pressure cuff, and the method is increasingly used in clinical trials. The mechanisms behind RIC are not yet fully understood, but the cardioprotective effects are believed to be caused by neural and humoral signaling cascades as well as systemic anti-inflammatory effects resulting in a cytoprotective state. In addition, RIC has been shown to reduce thrombus formation. Since activation of platelets and the coagulation system are fundamental in thrombus formation and degradation, another possible mechanism of the described effects of RIC could be a result from effect on arterial thrombus formation.

The vast majority of experimental and clinical studies have utilized RIC as single-occasion treatment (i.e. 3 or 4 bouts of short limb ischemia conducted once). However, experimental studies have recently suggested that repeated RIC treatment may infer further beneficial effects. Repeated RIC application has been shown to improve endothelial function and modify leukocyte adhesion in healthy volunteers. In a rat model of myocardial infarction, RIC repeated daily for 28 days after infarction reduced adverse ventricular remodeling and improved survival. Consequently, two on-going clinical trials (clinicaltrials.gov: DREAM study NCT01664611 and CRIC-RCT study NCT01817114) are investigating the effect of repeated RIC on LVEF function in patients with reduced ventricular function after an acute coronary event. Another study investigates the effect of repeated RIC on patients with severe heart failure and left ventricular assist device (IMPULSE study NCT02044471).

So far, the effect of RIC on patients suffering from stable chronic ischemic heart failure is unknown. Furthermore, no registered studies have evaluated the effect of long-term RIC given as additive treatment to the standard medical therapy in patients with chronic ischemic heart failure.

Hypothesis

• We hypothesize, that the combination of anti-remodelling and anti-inflammatory properties together with improved endothelial function induced by repetitive RIC treatment translate into improved left ventricular function and better physical performance in subjects with CHF.

Purpose

* To determine whether RIC applied on a daily basis for 4 weeks improves left ventricular function as assessed by cardiac magnetic resonance imaging (MRI) in subjects with CHF.
* To investigate whether RIC applied on a daily basis for 4 weeks improves muscle strength, cardiopulmonary exercise capacity and thrombocyte function, and changes blood biomarker levels of inflammation and heart failure in subjects with CHF.
* To investigate whether the above-mentioned measurements differ between patients with CHF and matched subjects after RIC applied on a daily basis for 4 weeks.

Perspectives The present study will elucidate whether long-term RIC treatment induces beneficial effects in subjects with and without chronic ischemic heart failure in terms of improved left ventricular contractile function and exercise capacity, and whether long-term RIC treatment induces systemic anti-inflammatory effects in these subjects. Moreover, we find that the study can uncover some of the mechanisms behind RIC and thus potentially optimize future treatment for patients suffering, or at risk, from ischemic heart diseases.

ELIGIBILITY:
Group 1 (Chronic heart failure patients):

Inclusion Criteria:

* >18 years of age
* Able to understand the written patient information and to give informed consent
* Chronic congestive ischemic heart failure
* Left ventricular ejection fraction ≤45%
* New York Heart Association functional class I-III

Exclusion Criteria:

* Recent cardiovascular hospitalization (within last 30 days) • Strenuous exercise within 72 hours of either study visits
* Intake of caffeine within 24 hours of either study visit
* Intake of alcohol within 24 hours of either study visit
* Patients with permanent atrial fibrillation • Patients with diabetes mellitus
* Patients with peripheral neuropathy
* Patients in dialysis treatment
* Contraindication for Magnetic Resonance Imaging examination (e.g. metal implants including Cardiac Resynchronisation Therapy devices and other pacemakers or defibrillators) precluding Magnetic Resonance Imaging
* Other concomitant disease or treatment that according to the investigator's assessment makes the patient unsuitable for study participation.

Group 2 (Volunteers without ischemic heart disease):

Inclusion criteria:

* >18 years of age
* Able to understand the written patient information and to give informed consent
* Left ventricular ejection fraction >45%

Exclusion criteria:

* Recent cardiovascular hospitalization (within last 30 days)
* Intake of acetylsalicylic acid or non-steroidal anti-inflammatory drug medication within 7 days of either study visit
* Strenuous exercise within 72 hours of either study visit
* Intake of caffeine within 24 hours of either study visit
* Intake of alcohol within 24 hours of either study visit
* Patients with ischemic heart disease
* Patients with diabetes mellitus
* Patients with peripheral neuropathy
* Patients in dialysis treatment
* Patients in treatment with Vitamin K-antagonists, adenosine diphosphate-receptor-inhibitor, oral anticoagulants or dipyridamol.
* Conditions contraindicating short term cessation of acetylsalicylic acid and/or non-steroidal anti-inflammatory drug intake
* Contraindication for Magnetic Resonance Imaging examination (e.g. metal implants) precluding Magnetic Resonance Imaging
* Other concomitant disease or treatment that according to the investigator's assessment makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction assessed by MRI | 28±4 days

SECONDARY OUTCOMES:
Global and regional myocardial function by strain analysis assessed by MRI | 28±4 days
Left ventricular mass and end-diastolic volume assessed by MRI | 28±4 days
Cardiac output assessed by MRI | 28±4 days
Cardiopulmonary exercise capacity assessed by staged exercise bicycle test and leg extension power rig test | 28±4 days
Serology markers for heart failure | 28±4 days
Serology inflammatory markers | 28±4 days

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Bøtker, Prof., Study Director — Department of Cardiology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital Skejby, Aarhus N, Dk-8200 Aarhus N, Denmark